CLINICAL TRIAL: NCT05540756
Title: Single-center, Observational Pilot Study on the Use of Intraoperative Neurophysiological Monitoring in Spinal Cord Stimulator Trials
Brief Title: Study on the Use of Intraoperative Neurophysiological Monitoring in Spinal Cord Stimulator Trials
Acronym: SCS-Monitor
Status: Withdrawn | Type: Observational
Why Stopped: lack of resources
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB22-0275
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Pain, Chronic; Lumbar Radiculopathy; SCS
Keywords: Spinal Cord Stimulator; Neuromonitoring; Lumbar radiculopathy; ELECTROMYOGRAPHY; Lumbar Pain; Muscle Action Potential; Intraoperative Neurophysiological Monitoring
MeSH Terms: conditions — Chronic Pain; Radiculopathy; Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SCS: Patients undergoing a spinal cord stimulator trial who is planning to have intraoperative neuromonitoring performed during the procedure

SUMMARY:
This is an observational pilot study. The spinal cord stimulator (SCS) procedure and neuromonitoring device is not under investigation. Neuromonitoring is typically performed on this patient population receiving SCS trials here. This study is collecting the data that is transmitted into EPIC from the device that is being collected as part of the patients standard of care. This study will specifically look at Boston Scientific SCS trials as those are the majority of SCS devices that are used here at this medical center

Primary Objective - To evaluate the difference between observed intraoperative neuromonitoring readings and patient reported coverage for spinal cord stimulator trials and

Secondary Objective(s) -

1. To evaluate the safety and tolerability of intraoperative neuromonitoring during spinal cord stimulator trials and via documented adverse events and patient elicited feedback on follow up questionnaires.
2. Patient satisfaction using PGIC from one week to 6-months post procedure
3. Change in pain intensity using NRS from baseline to 6-months post procedure

This study will follow subjects in conjunction with thier standard of care SCS clinic visits. This includes the one week wound check at the pain clinic and then a 2 week end of study phone call.

DETAILED DESCRIPTION:
Spinal cord stimulation (SCS) is a neuromodulation procedure that utilizes electrical stimulation via electrodes on the spinal cord for management of various chronic pain states. The most common indications for SCS placement include refractory neuropathic pain, complex regional pain syndromes (CRPS), post-laminectomy/failed back surgery syndrome, and ischemic limb pain related to peripheral vascular disease.1 Upon placing the percutaneous leads in the epidural space, the electrodes or the leads are activated with electrical currents and the patient is asked to report area of paresthesia in response to stimulation.

1. Hypothesis This study hypothesizes that one will be able to use percutaneous SCS leads and be able to properly map the dermatomal overlap with the myotomes recorded during the procedure using CMAP.
2. Objectives

Primary Objective - To evaluate the difference between observed intraoperative neuromonitoring readings and patient reported coverage for spinal cord stimulator trials and

Secondary Objective(s) -

1. To evaluate the safety and tolerability of intraoperative neuromonitoring during spinal cord stimulator trials and via documented adverse events and patient elicited feedback on follow up questionnaires.
2. Patient satisfaction using PGIC from one week to 6-months post procedure
3. Change in pain intensity using NRS from baseline to 6-months post procedure

Primary Study Endpoints The primary study endpoints will be the comparison between intraoperative neuromonitoring readings and patient reported coverage for spinal cord stimulator trials. This study will collect asleep tonic and sub-perception burst waveforms, as well as awake tonic and sub-perception burst waveforms. Also collected will be self-reported subject pain coverage with the subject awake and conversant.

2.5 Secondary Study Endpoints To evaluate the safety and tolerability of intraoperative neuromonitoring during spinal cord stimulator trials via documented adverse events and patient elicited feedback via NSR and PGIC.

SCS Neuromonitoring:

Subjects will be seen on the day of their procedure in the preoperative holding area. Once consent has been given, the patient will be taken to the OR and attached to monitors.

Once the subject is sedated, the IONM specialist will place subdermal needle electrodes in various muscle groups and begin testing to obtain baseline measurements. The muscle groups that will be monitored bilaterally are as follows: upper and lower intercostals, upper and lower abdomen, iliopsoas, vastus lateralis, biceps femoris, tibialis anterior, and gastrocnemius. Transcranial electrical stimulation electrodes will also be placed in the scalp with the patient mildly anesthetized to measure SSEPs and MEPs. Once IONM baselines are obtained, SCS leads will be placed.

Testing will begin with IONM with the patient under sedation. Intraoperatively, this study will employ the use of CMAP. After lead placement, the contacts of each lead will be activated with a sub-perception burst waveform and a tonic waveform. The study team will record the parameters and IONM response with the patients under sedation. Once confirmed with the IONM team, the anesthesia team will awaken the patient and cease sedation. With the patient awake, the coordinator will test the same regions while activating the same electrodes with the patient self-reporting their perceived areas of paresthesia. This will be done by asking the subject to confirm that the region being stimulated covers their region of pain.

Subjects will undergo the SCS trial as part of their standard of care and will be seen for follow-up 1 week post-trial, during which the leads will be pulled.

The patient will undergo SCS implant and be admitted for 24-hour postoperative observation. All follow-up visits and SCS procedures are part of standard of care.

Sequence and Duration of all Study Periods Total length for participation in this study is up to 2 weeks

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Lumbar Radiculopathy
* Expected to receive a Spinal Cord Stimulator trial at at the university of Chicago Medical Center

Exclusion Criteria:

* Subject is part of a vulnerable population.
* Cannot consent for themselves

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a SCS trial as part of thier standard of care who are diagnosed with lumbar radiculopathy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-12-10 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Spinal Cord Stimulator (SCS) Coverage | 2 Weeks
  Compare SCS coverage between intraoperative neuromonitoring readings and subject self-report. By testing 18 different muscle groups and then asking the subject to self-report the same muscle groups after they are awake.

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) | 2 Weeks
  Change in pain intensity using NRS from baseline to 2 weeks post procedure. NRS is an 11-point scale where 0 means no pain and 10 means the worst pain imaginable.
Patient Global Impression of Change (PGIC) | 2 Weeks
  Patient satisfaction using PGIC from baseline to 2 weeks post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Anitescu, MD PHD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States